CLINICAL TRIAL: NCT00180284
Title: SITELINE 2 Polyurethane Clinical Investigation
Brief Title: SITELINE 2 Polyurethane
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Clinicals0009
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2011-09-29 (Estimated); Status verified 2011-09

CONDITIONS: Bradycardia
Keywords: Pacemaker leads; Electrodes, implantable; Cardiac pacing, aritificial
MeSH Terms: conditions — Bradycardia

INTERVENTIONS:
Device: SITELINE 2 Polyurethane (pacing lead) — SITELINE 2 Polyurethane (pacing lead)

SUMMARY:
The SITELINE 2 Polyurethane Clinical Investigation analyzed the safety and electrical performance of the SITELINE 2 Polyurethane pacing lead.

DETAILED DESCRIPTION:
This was a prospective, single-arm, multi-center U.S. clinical investigation, designed to demonstrate the safety and effectiveness of the SITELINE 2 Polyurethane extendable, retractable pacing lead in humans

ELIGIBILITY:
Inclusion Criteria:

* Patients indicated for dual chamber pulse generator implant, where the pulse generator is capable of meeting the requirements of this investigational protocol
* Patients selected must have the study lead as the initial implant of a permanent pacing lead in both the right atrium and the right ventricle
* Age 18 or above, or of legal age to give informed consent specific to state and national law
* Willing and capable of undergoing a device implant and participating in all testing associated with this clinical investigation
* Available for follow-up at an approved clinical investigational center, at the protocol-defined intervals
* A life expectancy of more than 180 days

Exclusion Criteria:

* Have or who are likely to receive a mechanical tricuspid valve during the course of the clinical investigation
* Have surgically uncorrected primary valvular heart disease
* Have an atrial tachyarrhythmia that is permanent (i.e., does not terminate spontaneously and cannot be terminated with medical intervention) or persistent (i.e., can be terminated with medical intervention, but does not terminate spontaneously)
* Requiring ICD therapy
* Have a hypersensitivity to a nominal single dose of 1.0 mg (0.5 mg per electrode) of dexamethasone acetate drug
* Enrolled in any concurrent study, including drug investigation, without Guidant written approval, that may confound the results of this study
* Women who are pregnant or plan to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2004-11; Primary Completion 2005-05 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Pacing voltage threshold at 3 Months | 3 months
Pacing impedance at 3 Months | 3 months
Sensed amplitude at 3 Months | 3 months
Lead complication-free rate up to 3 Months | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple Locations in the United States, Saint Paul, Minnesota, United States